CLINICAL TRIAL: NCT05166122
Title: Implementation of an Integrated System of Artificial Intelligence and Referral Tracking for Real-time Diabetic Retinopathy Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Health Systems Research Institute,Thailand (Other Government); Google LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 64077
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Retinopathy; Artificial Intelligence; Screening
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI workflow (Active Comparator): In AI work flow, patients will be screened by taking normal retinal images and all images will be assessed for the severity of diabetic retinopathy by a computerized artificial intelligence system immediately after the photograph is taken via the Internet and retinal images will be sent to the retinal ophthalmologist for overreading.
  Interventions: Diagnostic Test: Artificial Intelligence
- Manual workflow (No Intervention): Volunteers who have been screened by manual workflow will be screened by imaging the retina and image that are not normal will be sent to assess the severity of diabetic retinopathy by specialist staff.

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence — Introduction of digitized system with an AI tool to detect and intrepret the severity of diabetic retinopathy and presence of diabetic macular edema in screening for diabetes patients
  Arms: AI workflow

SUMMARY:
This research study aims to bring an artificial intelligence system to screen for diabetic retinopathy (DR) along with referral tracking systems to the screening unit in Uthai Hospital in Phra Nakhon Sri Ayutthaya to assess the effectiveness of screening and follow-up of patients referred to Phra Nakhon Sri Ayutthaya Hospital. It will be compared with the existing screening system and follow up with regular referral by personnel

DETAILED DESCRIPTION:
Diabetic retinopathy is the most common ocular complication in people with diabetes. It is a leading cause of vision loss and blindness in people aged 20-64 years around the world because in the early stages of the disease there is no warning, causing the patients to be unaware. If the blood sugar content is allowed to increase, severe diabetic retinopathy can occur leading to blindness.

The incidence of diabetic retinopathy in diabetic patients tends to increase with the duration of diabetes. And according to the age of the patient, it was found that within 20 years, patients with diabetes type 1 with diabetic retinopathy is about 99% and diabetes type 2 with diabetic retinopathy is about 60%.

Screening for diabetic retinopathy is accepted and performed in health systems around the world. Evidence shows that screening can reduce blindness(1-3). Thailand uses the percentage of diabetic patients who have been eye tested. It is one of the indicators of service quality of the Eye Health District of the Ministry of Public Health. Screening for diabetic retinopathy using the retinal imaging method is cost-effective. It provides diabetic patients in distant places access to screening, such as bringing a mobile retina camera to take pictures in the community in conjunction with the use of teleophthalmology technology in screening(4-6). But according to a report by the Ministry of Public Health in the HDC system in 2015-2017, it was found that only 40% of the patients who were screened for diabetic retinopathy had not reached the 60% target.

In 2016, Rajavithi Hospital, in collaboration with researchers in Google Health, assessed the use of artificial intelligence to read retina images of diabetic patients in all 13 health districts of Thailand. It found that the artificial intelligence system was able to identify patients for referral to ophthalmologists (moderate non-proliferative diabetic retinopathy [NPDR]) with 95% sensitivity and 96% specificity, which is 73% higher than screening personnel specificity 98%.

From thereon, a prospective study with the introduction of artificial intelligence system was conducted to screen real patients in the project titled "Thailand-Google Prospective, Real-World Deployment of Artificial Intelligence for Diabetic Retinopathy Screening" (THAIGER) (NCT TCTR 20190902002) in 2018 to 2020 to assess the feasibility, including obstacles to implementing an intelligence-based screening process. The project integrated AI into the nation-wide screening system of the country. By conducting research in the primary care facilities, Rajavithi Hospital and 9 community hospitals in Pathum Thani Province and Chiang Mai, the diabetic patients in the THAIGER project received the results of reading images by artificial intelligence in real time. However, it was found that of the patients who were referred, very few actually went to see a doctor. There are also images that were unreadable (ungradable) by the artificial intelligence. And the artificial intelligence used in THAIGER has not yet been fully integrated into the screening system, including with a patient tracking system.

This research study aims to bring an artificial intelligence system to screen for diabetic retinopathy (DR) along with referral tracking systems to the screening unit in Uthai Hospital in Phra Nakhon Sri Ayutthaya to assess the effectiveness of screening and follow-up of patients referred to Phra Nakhon Sri Ayutthaya Hospital. It will be compared with the existing screening system and follow up with regular referral by personnel.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over.
* Patients who have been screened for diabetic retinopathy at Uthai Hospital Phra Nakhon Sri Ayutthaya Province that can refer patients to Phra Nakhon Sri Ayutthaya Hospital to see an ophthalmologist
* People with diabetes who are listed on the civil registry
* Able to take pictures of the retina at least 1 eye.

Exclusion Criteria:

* Being a patient in a community hospital with an in-house ophthalmologist
* Patients who were previously diagnosed for the following conditions / diseases: retinal edema, diabetic retinopathy (NPDR, PDR). The retina is affected by radiation (Radiation retinopathy) or retinal vein blockage (RVO).
* Past history of laser retinal treatment or retinal surgery
* Having other eye diseases (non-diabetic retinopathy) that requires referral to an ophthalmologist.
* Inability to take pictures of the retina (for any reason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Referral adherence | 6 months
  Total number of patients who completed referral visit in each arm (ie, presented to tertiary eye care center)

SECONDARY OUTCOMES:
User trust and acceptability | 6 months
  Assessment of staff satisfaction with workflows and patient experience in each arm
Screening throughput | Compare time unit of 1 day for each arm
  Assess the number of patients who successfully completed screening in a given day in the AI versus manual arm
Assess AI performance | 6 months
  Confirm sensitivity and specificity of AI reading as demonstrated in previous prospective study (THAIGER, TCTR20190902002)

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chotcomwongse P, Ruamviboonsuk P, Karavapitayakul C, Thongthong K, Amornpetchsathaporn A, Chainakul M, Triprachanath M, Lerdpanyawattananukul E, Arjkongharn N, Ruamviboonsuk V, Vongsa N, Pakaymaskul P, Waiwaree T, Ruampunpong H, Tiwari R, Tangcharoensathien V. Transforming Non-Digital, Clinical Workflows to Detect and Track Vision-Threatening Diabetic Retinopathy via a Digital Platform Integrating Artificial Intelligence: Implementation Research. Ophthalmol Ther. 2025 Feb;14(2):447-460. doi: 10.1007/s40123-024-01086-8. Epub 2025 Jan 10. PMID 39792334